CLINICAL TRIAL: NCT02605967
Title: A Phase II, Open-label, Randomized Controlled Study of PDR001 in Patients With Moderately Differentiated/Undifferentiated Locally Advanced Recurrent or Metastatic Nasopharyngeal Carcinoma Who Progressed on Standard Treatment
Brief Title: Safety and Efficacy Study of PDR001 in Patients With Recurrent or Metastatic Nasopharyngeal Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CPDR001X2201; 2015-000454-38 (EudraCT Number)
Record Dates: First submitted 2015-10-15; First posted 2015-11-17 (Estimated); Results first posted 2021-08-12 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-01

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: PDR001; nasopharyngeal cancer; moderately differentiated/undifferentiated; locally advanced; recurrent or metastatic NPC; after first- line platinum-based therapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma; Nasopharyngeal Neoplasms; Disorders of Sex Development; Recurrence | interventions — spartalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Spartalizumab 400 mg Q4W (Experimental): anti-PD1 humanized monoclonal antibody. Participants treated with spartalizumab who remained on spartalizumab
  Interventions: Drug: Spartalizumab
- Chemotherapy (Active Comparator): commonly used chemotherapy as per investigator's choice
  Interventions: Drug: Investigator choice of chemotherapy

INTERVENTIONS:
Drug: Spartalizumab — Spartalizumab was administered via intravenous infusion at a dose of 400 mg every 4 weeks (Q4W). Spartalizumab is a humanized anti-PD-1 IgG4 antibody which blocks the binding of PD1 to its ligands PD-L1 and PD-L2.
  Other Names: PDR001
  Arms: Spartalizumab 400 mg Q4W
Drug: Investigator choice of chemotherapy — Commonly used chemotherapy as per investigator's choice. The dose and route of administration was the one described in each drug's label.
  Arms: Chemotherapy

SUMMARY:
The purpose of this randomized controlled Phase II study is to assess the efficacy of PDR001 versus investigator's choice of chemotherapy in patients with advanced nasopharyngeal carcinoma (NPC).

By blocking the interaction between PD-1 and its ligands PD-L1 and PD-L2, PDR001 leads to the activation of a T-cell mediated antitumor immune response.

DETAILED DESCRIPTION:
This was an open-label, multi-center, randomized, and controlled Phase II study to evaluate the efficacy and safety of spartalizumab versus investigator's choice of treatment in subjects with moderately differentiated/undifferentiated locally advanced recurrent or metastatic NPC who progressed on or after first-line treatment.

Participants who met the inclusion/exclusion criteria were randomized in a 2:1 ratio to either investigational arm (spartalizumab) or control arm (commonly used chemotherapy as per investigator's choice). Participants treated with spartalizumab could continue treatment until confirmed progressive disease as per immune-related response criteria (irRC). Participants in the chemotherapy arm were allowed to crossover to spartalizumab if they had radiological progression as per Response Evaluation Criteria In Solid Tumors version 1.1 (RECIST v1.1) documented by an independent central review and the Investigator believed this was the best treatment option for the patient.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented non-keratinizing locally advanced recurrent or metastatic NPC.
* Must be resistant to platinum-based chemotherapy (defined as progression on or after platinum-based chemotherapy given in the recurrent/metastatic setting).
* May have received at least 1 prior therapy for recurrent or metastatic disease, up to 2 prior systemic therapies.
* An archival tumor specimen or newly obtained tumor sample may be submitted at screening/baseline (a fresh tumor sample is preferred), unless agreed differently between Novartis and the Investigator.
* At least 1 measurable lesion (as per RECIST v1.1) progressing or new since last anti-tumor therapy.
* Prior treated brain or meningeal metastases must be without MRI evidence of progression for at least 8 weeks and off systemic steroids for at least 2 weeks prior to screening/baseline.
* Patient must be willing to undergo testing for human immunodeficiency virus (HIV) if not tested within the past 6 months. If HIV+ positive, patient will be eligible if: his/ her CD4+ count ≥ 300/μL; his/her viral load is undetectable; he/she is currently receiving highly active antiretroviral therapy (HAART).

Exclusion Criteria:

* History of severe hypersensitivity reactions to other mAbs
* Active autoimmune disease or a documented history of autoimmune disease, except vitiligo or resolved asthma/atopy that is treated with broncho-dilators.
* Active HBV or HCV infections requiring therapy.
* Prior PD-1- or PD-L1-directed therapy or any therapeutic cancer vaccine.
* Patients receiving systemic treatment with any immunosuppressive medication.
* Use of any vaccines against infectious diseases (e.g. varicella, pneumococcus) within 4 weeks of initiation of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2016-04-20 (Actual); Primary Completion 2019-11-05 (Actual); Study Completion 2021-02-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (18):
- United States (4):
  - Northwest Georgia Oncology Center NWGA Onc - Carrollton, Marietta, Georgia
  - Karmanos Cancer Institute, Detroit, Michigan
  - NYU Laura and Isaac Perlmutter Cancer Center Laura & Isaac Perlmutter Ctr, New York, New York
  - Virginia Cancer Specialists, Fairfax, Virginia
- Novartis Investigative Site, Guangzhou, China
- France (2):
  - Novartis Investigative Site, Nice, Alpes Maritimes
  - Novartis Investigative Site, Villejuif, Villejuif
- Hong Kong (3):
  - Novartis Investigative Site, Hong Kong
  - Novartis Investigative Site, Kowloon
  - Novartis Investigative Site, Tuenmen
- Novartis Investigative Site, Singapore, Singapore
- Taiwan (4):
  - Novartis Investigative Site, Tainan, Taiwan ROC
  - Novartis Investigative Site, Kaohsiung City
  - Novartis Investigative Site, Taipei
  - Novartis Investigative Site, Taoyuan District
- Thailand (3):
  - Novartis Investigative Site, Songkhla, Hat Yai
  - Novartis Investigative Site, Bangkok
  - Novartis Investigative Site, Chiang Mai

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Even C, Wang HM, Li SH, Ngan RK, Dechaphunkul A, Zhang L, Yen CJ, Chan PC, Chakrabandhu S, Ma BBY, Tanasanvimon S, Lee VHF, Lou PJ, Li Z, Spira AI, Sukari A, Guigay J, McCune S, Gonzalez-Maffe J, Szpakowski S, Yao Y, Liang H, Mataraza J, Sechaud R, Manenti L, Lim DW. Phase II, Randomized Study of Spartalizumab (PDR001), an Anti-PD-1 Antibody, versus Chemotherapy in Patients with Recurrent/Metastatic Nasopharyngeal Cancer. Clin Cancer Res. 2021 Dec 1;27(23):6413-6423. doi: 10.1158/1078-0432.CCR-21-0822. Epub 2021 Aug 25. PMID 34433653

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in 19 investigative sites in 7 countries.
Pre-assignment Details: The screening period began once patients had signed the study informed consent. All screening evaluations were performed as closely as possible to the beginning of treatment and never more than 4 weeks before the beginning of the study treatment. After screening, the treatment period started on Cycle 1 Day 1.
Period: Overall Study
Arm/Group | Spartalizumab 400 mg Q4W | Chemotherapy
Started (All participants to whom study treatment was assigned by randomization) | 82 | 40
Safety Set (All participants who received at least one dose of study medication and had at least one valid post-screening/post-baseline safety assessment.) | 82 | 39
Crossover to Spartalizumab (Participants in Chemotherapy arm were allowed to crossover to spartalizumab treatment if they had radiological progression as per RECIST v1.1 by independent central review.) | 0 | 27
Completed | 0 | 0
Not Completed | 82 | 40
Not completed — subject / guardian decision | 1 | 2
Not completed — Physician Decision | 10 | 1
Not completed — Death | 4 | 2
Not completed — Adverse Event | 1 | 0
Not completed — progressive disease | 66 | 35

BASELINE CHARACTERISTICS:
Population: There were 122 participants in this trial. Of the 40 subjects from the chemotherapy arm, 25 subjects crossed over to receive spartalizumab.
Groups:
- Total: Total of all reporting groups
Arm/Group | Spartalizumab 400 mg Q4W | Chemotherapy | Total
Number analyzed (Participants) | 82 | 40 | 122
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.1 (11.54) | 50.5 (12.32) | 50.9 (11.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 7 | 21
  Male | 68 | 33 | 101
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 12 | 2 | 14
  Black | 0 | 1 | 1
  Asian | 70 | 37 | 107

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) as Per RECIST v 1.1 Using Central Assessment - Number of Participants With Progression or Death
Description: PFS is the time from the date of randomization to the date of event defined as the first documented confirmed progression or death due to any cause. If a patient has not had an event, progression-free survival is censored at the date of last adequate tumor assessment.
  Tumor response was based on central review of tumor scan and the assessment criteria was Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1). Progressive disease is at least a 20% increase in the sum of diameter of all measured target lesions, taking as reference the smallest sum of diameter of all target lesions recorded at or after baseline. Number of participants in each category (progression, death, censored) is reported in this record.
Time Frame: From randomization up to maximum 3.3 years
Population: All participants to whom study treatment was assigned by randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Spartalizumab 400 mg Q4W | Chemotherapy
Number analyzed (Participants) | 82 | 40
Participants
  number of progression | 62 | 32
  number of deaths | 3 | 1
  number of censored | 17 | 7

2. Primary Outcome: Progression-free Survival (PFS) as Per RECIST v 1.1 Using Central Assessment - Median PFS
Description: PFS is the time from the date of randomization to the date of event defined as the first documented confirmed progression or death due to any cause. If a patient has not had an event, progression-free survival is censored at the date of last adequate tumor assessment.
  Tumor response was based on central review of tumor scan and the assessment criteria was Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1). Progressive disease is at least a 20% increase in the sum of diameter of all measured target lesions, taking as reference the smallest sum of diameter of all target lesions recorded at or after baseline.
Time Frame: From randomization up to maximum 3.3 years
Population: All participants to whom study treatment was assigned by randomization.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Spartalizumab 400 mg Q4W | Chemotherapy
Number analyzed (Participants) | 82 | 40
months | 1.9 [1.8 to 2.9] | 5.6 [3.7 to 9.2]

3. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) is defined as the time from date of randomization to date of death due to any cause. If a patient is not known to have died, survival is censored at the date of last known date the patient was alive.
Time Frame: From randomization up to maximum 4.8 years.
Population: All participants to whom study treatment was assigned by randomization.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Spartalizumab 400 mg Q4W | Chemotherapy
Number analyzed (Participants) | 82 | 40
months | 20.1 [13.6 to 25.5] | 16.0 [8.8 to 22.5]

4. Secondary Outcome: Overall Response Rate (ORR) as Per RECIST v 1.1
Description: ORR is defined as the percentage of participants with a best overall response of Complete Response (CR) or Partial Response (PR). Tumor response was based on central review of overall lesion response according to RECIST 1.1.
  For RECIST v1.1, CR=Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm; PR= At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: From randomization up to maximum 3.3 years
Population: All participants to whom study treatment was assigned by randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Spartalizumab 400 mg Q4W | Chemotherapy
Number analyzed (Participants) | 82 | 40
Participants | 15 | 13

5. Secondary Outcome: Duration of Response (DOR) as Per RECIST v 1.1
Description: DOR only applies to subjects for whom best overall response is complete response (CR) or partial response (PR) based on central review of overall lesion response according to RECIST 1.1. DOR is defined as the time between the date of first documented response (confirmed CR or confirmed PR) and the date of first documented disease progression or death due to underlying cancer. If a patient not had an event, duration was censored at the date of last adequate tumor assessment.
Time Frame: From randomization up to maximum 3.3 years
Population: All participants for whom best overall response is complete response (CR) or partial response (PR) as per RECIST 1.1 based on central review.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Spartalizumab 400 mg Q4W | Chemotherapy
Number analyzed (Participants) | 15 | 13
months | 10.2 [7.4 to NA] — Not estimable due to insufficient number of participants with events. | 5.7 [3.7 to 7.4]

6. Secondary Outcome: Time to Progression (TTP) as Per RECIST v 1.1
Description: TTP is defined as time from date of randomization to the date of event defined as the first documented progression or death due to underlying cancer. If a subject did not had an event, TTP was censored at the date of last adequate tumor assessment.
  Tumor response was based on central review of tumor scan and the assessment criteria was RECIST v1.1. Progressive disease is at least a 20% increase in the sum of diameter of all measured target lesions, taking as reference the smallest sum of diameter of all target lesions recorded at or after baseline.
Time Frame: From randomization up to maximum 3.3 years
Population: All participants to whom study treatment was assigned by randomization.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Spartalizumab 400 mg Q4W | Chemotherapy
Number analyzed (Participants) | 82 | 40
months | 1.9 [1.8 to 2.9] | 5.6 [3.7 to 9.3]

7. Secondary Outcome: Immune-related Progression-free Survival (irPFS) as Per irRC
Description: irPFS is the time from the date of randomization to the date of event defined as the first documented progression or death due to any cause. If a patient has not had an event, progression-free survival is censored at the date of last adequate tumor assessment.
  Tumor response was based on central review of tumor scan and the assessment criteria was immune-related Response Criteria (irRC). Immune-related progressive disease is at least a 20% increase in the sum of diameters of all measured target lesions including new measurable lesions.
Time Frame: From randomization up to maximum 3.3 years
Population: All participants to whom study treatment was assigned by randomization to spartalizumab. For the chemotherapy arm, tumor scans for efficacy assessment as per irRC were not planned.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Spartalizumab 400 mg Q4W | Chemotherapy
Number analyzed (Participants) | 82 | 0
months | 1.9 [1.8 to 3.6] |

8. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) of Spartalizumab
Description: Pharmacokinetic (PK) parameters were calculated based on spartalizumab serum concentrations by using non-compartmental methods. Cmax is defined as the maximum (peak) observed serum concentration following a dose.
Time Frame: pre-dose, 1, 24, 168, 336 and 672 hours post spartalizumab dose on Cycle 1 and Cycle 3. The duration of one cycle was 28 days.
Population: All participants who had at least one dose of spartalizumab and had at least one evaluable concentration measurement of spartalizumab. PK samples were only collected in participants to whom spartalizumab was assigned by randomization.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Spartalizumab 400 mg Q4W
Number analyzed (Participants) | 82
ug/mL
  Cycle 1: number analyzed (Participants) | 78
  Cycle 1 | 116 (21.9)
  Cycle 3: number analyzed (Participants) | 47
  Cycle 3 | 149 (25.8)

9. Secondary Outcome: Time to Reach Maximum Serum Concentration (Tmax) of Spartalizumab
Description: Pharmacokinetic (PK) parameters were calculated based on spartalizumab serum concentrations by using non-compartmental methods. Tmax is defined as the time to reach maximum (peak) serum concentration following a dose. Actual recorded sampling times were considered for the calculations.
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Median (Full Range); unit: hours
Arm/Group | Spartalizumab 400 mg Q4W
Number analyzed (Participants) | 82
hours
  Cycle 1: number analyzed (Participants) | 78
  Cycle 1 | 1.57 [0.58 to 3.17]
  Cycle 3: number analyzed (Participants) | 47
  Cycle 3 | 1.57 [1.00 to 14.9]

10. Secondary Outcome: Area Under the Serum Concentration-time Curve From Time Zero to the End of the Dosing Interval Tau (AUCtau) of Spartalizumab
Description: Pharmacokinetic (PK) parameters were calculated based on spartalizumab serum concentrations by using non-compartmental methods. The linear trapezoidal method was used for AUC calculation. The duration of the dosing interval (tau) was 28 days.
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*ug/mL
Arm/Group | Spartalizumab 400 mg Q4W
Number analyzed (Participants) | 82
day*ug/mL
  Cycle 1: number analyzed (Participants) | 73
  Cycle 1 | 1340 (25.8)
  Cycle 3: number analyzed (Participants) | 39
  Cycle 3 | 2260 (30.6)

11. Secondary Outcome: Area Under the Serum Concentration-time Curve From Time Zero to Infinity (AUCinf) of Spartalizumab
Description: Pharmacokinetic (PK) parameters were calculated based on spartalizumab serum concentrations by using non-compartmental methods. The linear trapezoidal method was used for AUC calculation. The extrapolation of AUC to infinity could be calculated if the percentage of area extrapolated was less than 20% and the regression analysis of the terminal serum elimination phase met a pre-defined criteria of goodness of fit.
Time Frame: as for outcome 8
Population: All participants who had at least one dose of spartalizumab and the extrapolation of AUC to infinity could be calculated as described in the description of the endpoint. PK samples were only collected in participants to whom spartalizumab was assigned by randomization.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*ug/mL
Arm/Group | Spartalizumab 400 mg Q4W
Number analyzed (Participants) | 7
day*ug/mL
  Cycle 1: number analyzed (Participants) | 6
  Cycle 1 | 1180 (23.9)
  Cycle 3: number analyzed (Participants) | 2
  Cycle 3 | 1090 (84.8)

12. Secondary Outcome: Accumulation Ratio (Racc) of Spartalizumab
Description: Pharmacokinetic (PK) parameters were calculated based on spartalizumab serum concentrations by using non-compartmental methods. Racc was calculated as the ratio between AUCtau Cycle 3 and AUCtau Cycle 1.
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Spartalizumab 400 mg Q4W
Number analyzed (Participants) | 39
ratio | 1.61 (19.6)

13. Secondary Outcome: Terminal Elimination Half-life (T1/2) of Spartalizumab
Description: Pharmacokinetic (PK) parameters were calculated based on spartalizumab serum concentrations by using non-compartmental methods. Elimination half-life (T1/2) values were calculated as 0.693/terminal elimination rate constant.
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Median (Full Range); unit: days
Arm/Group | Spartalizumab 400 mg Q4W
Number analyzed (Participants) | 82
days
  Cycle 1: number analyzed (Participants) | 79
  Cycle 1 | 20.1 [7.35 to 41.5]
  Cycle 3: number analyzed (Participants) | 48
  Cycle 3 | 22.7 [5.29 to 48.9]

14. Secondary Outcome: Number of Participants With Anti-spartalizumab Antibodies
Description: Validated immunoassays were used for screening and confirmation of the presence of anti-spartalizumab antibodies (ADA, anti-drug antibodies) in serum. Number of participants with each ADA status is reported in this record.
Time Frame: Baseline (pre-dose on Cycle 1 Day 1) and post-baseline (assessed throughout the treatment up to maximum 655 days).
Population: All participants who had at least one dose of spartalizumab and had a determinant baseline immunogenicity (IG) sample and at least one determinant post-baseline IG sample. A determinant IG sample is neither ADA-inconclusive nor unevaluable. IG samples were only collected in participants to whom spartalizumab was assigned by randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Spartalizumab 400 mg Q4W
Number analyzed (Participants) | 72
Participants
  ADA-negative at baseline | 66
  ADA-positive at baseline | 6
  ADA-negative at post-baseline | 59
  ADA-positive at post-baseline (i.e. ADA incidence) | 9

15. Secondary Outcome: PD-L1 Percent Positive Tumor
Description: The expression of programmed cell death-ligand 1 (PD-L1) was measured in tumor samples by immunohistochemical methods. This record summarizes the PD-L1 positivity percentage in tumor samples.
Time Frame: Baseline (screening), Cycle 3 Day 1. The duration of one cycle was 28 days.
Population: All participants to whom study treatment was assigned by randomization to spartalizumab and had a valid assessment for the outcome measure. Biomarker samples were not collected in participants randomized to chemotherapy.
Measure: Median (Full Range); unit: PD-L1 positivity percentage
Units Other Than Participants: tumor samples
Arm/Group | Spartalizumab 400 mg Q4W
Number analyzed (Participants) | 78
Number analyzed (tumor samples) | 79
PD-L1 positivity percentage
  Baseline: number analyzed (tumor samples) | 78
  Baseline | 20.00 [0 to 100]
  Cycle 3 Day 1: number analyzed (Participants) | 1
  Cycle 3 Day 1: number analyzed (tumor samples) | 1
  Cycle 3 Day 1 | 90.00 [90.00 to 90.00]

16. Secondary Outcome: Percent Marker Area for CD8 Expression in Tumor Samples
Description: The expression of CD8 was measured in tumor samples by immunohistochemical methods. This record summarizes the percent marker area for CD8 expression in tumor samples.
Time Frame: Baseline (screening), Cycle 3 Day 1. The duration of one cycle was 28 days.
Population: as for outcome 15
Measure: Median (Full Range); unit: CD8 percent marker area
Units Other Than Participants: tumor samples
Arm/Group | Spartalizumab 400 mg Q4W
Number analyzed (Participants) | 78
Number analyzed (tumor samples) | 79
CD8 percent marker area
  Baseline: number analyzed (tumor samples) | 78
  Baseline | 4.23 [0.1 to 31.8]
  Cycle 3 Day 1: number analyzed (Participants) | 1
  Cycle 3 Day 1: number analyzed (tumor samples) | 1
  Cycle 3 Day 1 | 2.22 [2.22 to 2.22]

17. Secondary Outcome: TIL Count in Tumor Samples
Description: The count of tumor-infiltrating lymphocytes (TILs) was measured in baseline (screening) and post-baseline paired tumor samples by immunohistochemical methods. This record summarizes the TIL count in tumor samples.
Time Frame: Baseline (screening), Cycle 3 Day 1. The duration of one cycle was 28 days.
Population: All participants to whom study treatment was assigned by randomization to spartalizumab and had paired tumor biopsies. Biomarker samples were not collected in participants randomized to chemotherapy.
Measure: Number; unit: TILs
Arm/Group | Spartalizumab 400 mg Q4W
Number analyzed (Participants) | 1
TILs
  Baseline | 10
  Cycle 3 Day 1 | 15

18. Secondary Outcome: Fold Change From Baseline in IFN-gamma Levels in Plasma
Description: The levels of interferon-gamma (IFN-gamma) were measured in plasma samples by immunoassay methods. This record summarizes the fold change from baseline in IFN-gamma levels in plasma.
Time Frame: Baseline (pre-dose on Cycle 1 Day 1), Cycle 1 Day 15, Cycle 2 Day 15 and end of treatment (assessed up to maximum 4 years). The duration of one cycle was 28 days.
Population: All participants to whom study treatment was assigned by randomization to spartalizumab. Biomarker samples were not collected in participants randomized to chemotherapy.
Measure: Median (Full Range); unit: fold change
Arm/Group | Spartalizumab 400 mg Q4W
Number analyzed (Participants) | 82
fold change
  Cycle 1 Day 15: number analyzed (Participants) | 65
  Cycle 1 Day 15 | 1.53 [0.2 to 14.3]
  Cycle 2 Day 15: number analyzed (Participants) | 51
  Cycle 2 Day 15 | 1.31 [0.1 to 35.2]
  End of treatment: number analyzed (Participants) | 34
  End of treatment | 1.11 [0.1 to 3.8]

19. Secondary Outcome: Fold Change From Baseline in IL-6 Levels in Plasma
Description: The levels of interleukin-6 (IL-6) were measured in plasma samples by immunoassay methods. This record summarizes the fold change from baseline in IL-6 levels in plasma.
Time Frame: as for outcome 18
Population: as for outcome 18
Measure: Median (Full Range); unit: fold change
Arm/Group | Spartalizumab 400 mg Q4W
Number analyzed (Participants) | 82
fold change
  Cycle 1 Day 15: number analyzed (Participants) | 41
  Cycle 1 Day 15 | 1.10 [0.2 to 3.3]
  Cycle 2 Day 15: number analyzed (Participants) | 30
  Cycle 2 Day 15 | 1.35 [0.2 to 6.3]
  End of treatment: number analyzed (Participants) | 26
  End of treatment | 1.41 [0.2 to 7.7]

20. Secondary Outcome: Fold Change From Baseline in TNF-alfa Levels in Plasma
Description: The levels of tumor necrosis factor-alpha (TNF-alfa) were measured in plasma samples by immunoassay methods. This record summarizes the fold change from baseline in TNF-alfa levels in plasma.
Time Frame: as for outcome 18
Population: as for outcome 18
Measure: Median (Full Range); unit: fold change
Arm/Group | Spartalizumab 400 mg Q4W
Number analyzed (Participants) | 82
fold change
  Cycle 1 Day 15: number analyzed (Participants) | 73
  Cycle 1 Day 15 | 1.32 [0.4 to 2.2]
  Cycle 2 Day 15: number analyzed (Participants) | 62
  Cycle 2 Day 15 | 1.39 [0.3 to 3.1]
  End of treatment: number analyzed (Participants) | 45
  End of treatment | 1.67 [0.3 to 3.7]

21. Post Hoc Outcome: Progression-free Survival (PFS) as Per RECIST v 1.1 Using Central Assessment in Participants Who Crossed Over - Number of Participants With Progression or Death
Description: PFS is the time from the date of first dose of spartalizumab to the date of event defined as the first documented confirmed progression or death due to any cause. If a patient has not had an event, progression-free survival is censored at the date of last adequate tumor assessment.
  Tumor response was based on central review of tumor scan and the assessment criteria was Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1). Progressive disease is at least a 20% increase in the sum of diameter of all measured target lesions, taking as reference the smallest sum of diameter of all target lesions recorded at or after baseline. Number of participants in each category (progression, death, censored) is reported in this record.
Time Frame: From first dose of spartalizumab up to maximum 0.6 years
Population: All participants who crossed over from chemotherapy to spartalizumab.
Measure: Count of Participants; unit: Participants
Groups:
- Crossover to Spartalizumab: Patients treated with chemotherapy who crossed over to spartalizumab
Arm/Group | Crossover to Spartalizumab
Number analyzed (Participants) | 27
Participants
  number of progression | 20
  number of deaths | 5
  number of censored | 2

22. Post Hoc Outcome: Progression-free Survival (PFS) as Per RECIST v 1.1 Using Central Assessment in Participants Who Crossed Over - Median PFS
Description: PFS is the time from the date of first dose of spartalizumab to the date of event defined as the first documented confirmed progression or death due to any cause. If a patient has not had an event, progression-free survival is censored at the date of last adequate tumor assessment.
  Tumor response was based on central review of tumor scan and the assessment criteria was Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1). Progressive disease is at least a 20% increase in the sum of diameter of all measured target lesions, taking as reference the smallest sum of diameter of all target lesions recorded at or after baseline.
Time Frame: From first dose of spartalizumab up to maximum 0.6 years
Population: All participants who crossed over from chemotherapy to spartalizumab.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Crossover to Spartalizumab
Number analyzed (Participants) | 27
months | 1.7 [1.6 to 1.9]

23. Post Hoc Outcome: All Collected Deaths
Description: On-treatment deaths were collected from the start of treatment up to 30 days after study drug discontinuation, for a maximum duration of 4.0 years. Post-treatment deaths were collected after the on-treatment period (starting at day 31 after last dose of study treatment), up to 4.8 years.
  For the crossover patients, the deaths collected before crossing over are summarized in the chemotherapy arm and the deaths collected after the crossover are summarized in the crossover arm.
Time Frame: Up to 4.0 years (on-treatment deaths) and 4.8 years (all deaths).
Population: All participants to whom study treatment was assigned by randomization.
Measure: Number; unit: participants
Arm/Group | Spartalizumab 400 mg Q4W | Chemotherapy | Crossover to Spartalizumab
Number analyzed (Participants) | 82 | 40 | 27
participants
  Total Deaths | 48 | 9 | 19
  Deaths on-treatment | 5 | 3 | 3

ADVERSE EVENTS:
Time Frame: From first dose of study treatment up to 30 days after last dose (maximum 4.0 years).
Description: For the crossover patients, safety data collected before crossing over is summarized in the chemotherapy arm and safety data collected after the crossover is summarized in the crossover arm.
  The column 'all spartalizumab participants' summarizes the safety data of the 2 arms with spartalizumab dosing.
  AEs and mortality are assessed in the safety set that includes all patients who received at least 1 dose of study medication and had at least 1 valid post-screening/post-baseline safety assessment.
Groups:
- All Spartalizumab Participants: All participants who received at least one dose of spartalizumab
Arm/Group | Spartalizumab 400 mg Q4W | Chemotherapy | Crossover to Spartalizumab | All Spartalizumab Participants
All-Cause Mortality (participants affected / at risk) | 5/82 | 3/39 | 3/27 | 8/109
Serious Adverse Events (participants affected / at risk) | 28/82 | 15/39 | 12/27 | 40/109
Other Adverse Events (participants affected / at risk) | 76/82 | 37/39 | 25/27 | 101/109
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Spartalizumab 400 mg Q4W (N=82) | Chemotherapy (N=39) | Crossover to Spartalizumab (N=27) | All Spartalizumab Participants (N=109)
Anaemia (Blood and lymphatic system disorders) | 2 | 1 | 1 | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 4 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Normocytic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0 | 1
Papilloedema (Eye disorders) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1 | 2
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 1 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 2 | 1 | 2
Asthenia (General disorders) | 1 | 1 | 1 | 2
Fatigue (General disorders) | 0 | 1 | 1 | 1
Generalised oedema (General disorders) | 0 | 0 | 1 | 1
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0
Pain (General disorders) | 0 | 1 | 0 | 0
Peripheral swelling (General disorders) | 0 | 0 | 1 | 1
Pyrexia (General disorders) | 3 | 0 | 1 | 4
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 1 | 1
Hepatocellular injury (Hepatobiliary disorders) | 1 | 0 | 0 | 1
Brain abscess (Infections and infestations) | 0 | 1 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 1 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1 | 1 | 2
Sepsis (Infections and infestations) | 2 | 0 | 1 | 3
Septic shock (Infections and infestations) | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 1
Electrical burn (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 2 | 0 | 0 | 2
Bilirubin conjugated increased (Investigations) | 1 | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 1
Blood bilirubin unconjugated increased (Investigations) | 1 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0 | 1 | 3
Malnutrition (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 1
Diplegia (Nervous system disorders) | 1 | 0 | 0 | 1
Hemiparesis (Nervous system disorders) | 1 | 0 | 0 | 1
Spinal cord compression (Nervous system disorders) | 2 | 1 | 0 | 2
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 3
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Miscarriage of partner (Social circumstances) | 1 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Spartalizumab 400 mg Q4W (N=82) | Chemotherapy (N=39) | Crossover to Spartalizumab (N=27) | All Spartalizumab Participants (N=109)
Anaemia (Blood and lymphatic system disorders) | 19 | 19 | 6 | 25
Leukopenia (Blood and lymphatic system disorders) | 2 | 3 | 0 | 2
Lymphopenia (Blood and lymphatic system disorders) | 0 | 2 | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 12 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 3 | 0 | 1
Hypothyroidism (Endocrine disorders) | 10 | 2 | 3 | 13
Abdominal discomfort (Gastrointestinal disorders) | 0 | 2 | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 5 | 0 | 1 | 6
Abdominal pain (Gastrointestinal disorders) | 5 | 2 | 4 | 9
Abdominal pain upper (Gastrointestinal disorders) | 8 | 3 | 3 | 11
Constipation (Gastrointestinal disorders) | 13 | 7 | 3 | 16
Diarrhoea (Gastrointestinal disorders) | 5 | 5 | 1 | 6
Dry mouth (Gastrointestinal disorders) | 3 | 3 | 1 | 4
Dyspepsia (Gastrointestinal disorders) | 0 | 2 | 1 | 1
Dysphagia (Gastrointestinal disorders) | 5 | 1 | 0 | 5
Mouth ulceration (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 13 | 8 | 4 | 17
Oral pain (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 6 | 9 | 0 | 6
Vomiting (Gastrointestinal disorders) | 14 | 6 | 7 | 21
Asthenia (General disorders) | 11 | 2 | 1 | 12
Fatigue (General disorders) | 14 | 15 | 5 | 19
Malaise (General disorders) | 6 | 2 | 1 | 7
Oedema peripheral (General disorders) | 2 | 5 | 0 | 2
Peripheral swelling (General disorders) | 0 | 0 | 2 | 2
Pyrexia (General disorders) | 16 | 3 | 8 | 24
Swelling face (General disorders) | 0 | 3 | 1 | 1
Herpes zoster (Infections and infestations) | 3 | 2 | 0 | 3
Nasopharyngitis (Infections and infestations) | 3 | 2 | 0 | 3
Pneumonia (Infections and infestations) | 3 | 2 | 0 | 3
Sinusitis (Infections and infestations) | 1 | 2 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 9 | 2 | 1 | 10
Urinary tract infection (Infections and infestations) | 1 | 2 | 0 | 1
Alanine aminotransferase increased (Investigations) | 7 | 6 | 1 | 8
Aspartate aminotransferase increased (Investigations) | 15 | 7 | 2 | 17
Blood alkaline phosphatase increased (Investigations) | 4 | 1 | 2 | 6
Blood creatinine increased (Investigations) | 5 | 2 | 1 | 6
Blood thyroid stimulating hormone increased (Investigations) | 6 | 1 | 0 | 6
Lymphocyte count decreased (Investigations) | 3 | 2 | 1 | 4
Neutrophil count decreased (Investigations) | 1 | 2 | 0 | 1
Platelet count decreased (Investigations) | 1 | 7 | 2 | 3
Weight decreased (Investigations) | 9 | 5 | 0 | 9
White blood cell count decreased (Investigations) | 1 | 8 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 16 | 9 | 8 | 24
Dehydration (Metabolism and nutrition disorders) | 3 | 2 | 0 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 5 | 1 | 0 | 5
Hypoalbuminaemia (Metabolism and nutrition disorders) | 6 | 2 | 3 | 9
Hypokalaemia (Metabolism and nutrition disorders) | 5 | 13 | 4 | 9
Hypomagnesaemia (Metabolism and nutrition disorders) | 7 | 6 | 2 | 9
Hyponatraemia (Metabolism and nutrition disorders) | 14 | 6 | 4 | 18
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 2 | 5 | 14
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 6 | 4 | 13
Bone pain (Musculoskeletal and connective tissue disorders) | 4 | 2 | 1 | 5
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 4 | 3 | 0 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0 | 1
Dizziness (Nervous system disorders) | 5 | 1 | 3 | 8
Headache (Nervous system disorders) | 12 | 4 | 1 | 13
Hypoaesthesia (Nervous system disorders) | 4 | 5 | 2 | 6
Neuropathy peripheral (Nervous system disorders) | 3 | 5 | 2 | 5
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 4 | 0 | 0
Insomnia (Psychiatric disorders) | 9 | 3 | 3 | 12
Urinary retention (Renal and urinary disorders) | 0 | 0 | 2 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 17 | 12 | 1 | 18
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 0 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 | 3 | 3 | 15
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 10 | 3 | 0 | 10
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 1 | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 3 | 5
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 1 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 9 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 5 | 0 | 2 | 7
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 6 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 10 | 3 | 4 | 14
Rash (Skin and subcutaneous tissue disorders) | 15 | 6 | 1 | 16
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Hypertension (Vascular disorders) | 1 | 2 | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2019-06-24): https://cdn.clinicaltrials.gov/large-docs/67/NCT02605967/Prot_002.pdf
  • Statistical Analysis Plan (2021-03-23): https://cdn.clinicaltrials.gov/large-docs/67/NCT02605967/SAP_003.pdf